CLINICAL TRIAL: NCT06245018
Title: An Open, Dose Escalation and Extension Platform Trial to Evaluate the Safety, Pharmacological and Preliminary Efficacy of Human Induced Pluripotent Stem Cell Derived Natural Killer Cells (iNK) in Chinese Subjects With Solid Tumor
Brief Title: A Trial to Evaluate the Safety and Preliminary Efficacy of iNK in the Treatment of Subjects With Solid Tumor
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nuwacell Biotechnologies Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: iNK-1002
Record Dates: First submitted 2024-01-18; First posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor
Keywords: iNK
MeSH Terms: interventions — Ink

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- iNK Injection (Experimental): Cohort1:Low dose iNK injection; Cohort2:Mid dose iNK injection; Cohort3:High dose iNK injection;
  Interventions: Biological: iNK Injection

INTERVENTIONS:
Biological: iNK Injection — Subjects will receive about 4 cycles of iNK

SUMMARY:
This trial is to investigate the safety, efficacy of iNK in subjects with solid tumor. It is a dose escalation and extension trial.

DETAILED DESCRIPTION:
Solid tumor is a disease with high mortality rates. The aim of this trial is to investigate the safety, efficacy of iNK in subjects with solid tumor. It is a dose escalation and extension trial.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old.
2. Subjects with recurrent or metastatic solid tumors that cannot accept radical locoregional therapy;
3. Systemic standard treatment failed or cannot tolerate serious toxicity or lack of standard treatment.
4. Have 1 or more focus can be accessed according to RECIST 1.1
5. Eastern Cooperative Oncology Group(ECOG):0-1
6. Expected survival period over 3 months
7. Have acceptable organ function and the results of laboratory examination meet the request below:

   Hepatic Insufficiency (ALT) and Aspartate aminotransferase（AST）≤3xULN(upper limit of normal);Total Bilirubin≤3xULN；Creatinine≤3xULN；White blood cell count ≥3.0x10^9/L; Absolute Neutrophil Count≥1.0x10^9/L
8. Agree to contraception
9. Subjects who understand and voluntarily sign the Informed Consent Form（ICF)

Exclusion Criteria:

1. Central nervous system metastasis or meningeal metastasis with clinical symptoms；
2. With active infection during screening
3. Have serious or uncontrolled basic diseases;
4. Have continuous adverse event caused by previous anti-tumor therapy that might affect the evaluation of drug safety；
5. Accept anti-tumor therapy within 28 days before first injection;
6. Accept general anesthesia surgery or radiation therapy within 28 days before first injection;
7. Accept live vaccine or attenuated live vaccine within 28 days before first injection;
8. Allergy to known drug components;
9. Serous cavity effusion requiring clinical intervention；
10. Pregnancy or prepare to pregnant during the treatment;
11. Other situations that not suitable to participate into this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Event(AE) ，Serious Adverse Event(SAE)，Treatment Emergent Adverse Event（TEAE）and Treatment Related Adverse Event(TRAE) | From the date of initial infusion to a year after initial infusion
  Number of participants with treatment-related adverse events or serious adverse events as assessed by CTCAE v5.0
Dose-Limiting Toxicity(DLT) | 4 weeks after initial infusion
  Number of participants with Dose-limiting toxicity in 28 days after injection

SECONDARY OUTCOMES:
Objective Response Rate（ORR） | During the whole study
  Percentage of participants achieved Complete Response(CR) or Partial Response(PR)
Disease Control Rate（DCR） | From the date of initial infusion to a year after initial infusion
  Percentage of participants achieved Complete Response(CR) or Partial Response(PR) or Stable Disease(SD)
Duration Of Response（DOR） | First Injection to a year after Last Injection
  Duration for the first PR to the first Progressive Disease(PD)

IPD SHARING:
Plan to Share IPD: No